CLINICAL TRIAL: NCT01604707
Title: Medical Yoga for Patients With Stress-related Symptoms and Diagnoses in Primary Health Care - a Randomized Controlled Trial
Brief Title: Medical Yoga for Patients With Stress-related Symptoms and Diagnoses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Örebro County (Other)
Responsible Party: Principal Investigator, Elisabeth Westerdahl, PhD, Registered Physiotherapist, Region Örebro County
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MEDYOG 1
Record Dates: First submitted 2012-05-15; First posted 2012-05-24 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-10

CONDITIONS: Stress; Anxiety; Depression
Keywords: stress; anxiety; depression; quality of life
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): Standard care
- Medical Yoga (Experimental): Group training with medical yoga in primary health care.
  Interventions: Other: Medical Yoga

INTERVENTIONS:
Other: Medical Yoga — Patients were randomly allocated to a control group receiving standard care, or a yoga group treated with Medical yoga for 1 hour, once a week, over a 12-week period in addition to the standard care.
  Other Names: Medical Yoga group
  Arms: Medical Yoga

SUMMARY:
Background An increasing number of patients are suffering from stress-related symptoms and diseases. No scientific studies have examined the effects of Medical yoga on stress-related symptoms in patients in primary care. The purpose of this study was to evaluate Medical yoga treatment in patients with stress-related symptoms and diagnosis in primary health care.

Methods A randomized, controlled study was performed at a primary health care centre in Sweden from March to June 2011. Patients were randomly allocated to a control group receiving standard care, or a yoga group treated with Medical yoga for 1 hour, once a week, over a 12-week period in addition to the standard care. A total of 37 men and women, mean age 53±12 years, seeking care for stress-related symptoms at the primary health care centre were included and followed up after the 12-week study period. General stress level (measured using Perceived Stress Scale (PSS)), burnout (Shirom-Melamed Burnout Questionnaire (SMBQ)), anxiety and depression (Hospital Anxiety and Depression Scale (HADS)), insomnia severity (Insomnia Severity Index (ISI)), pain (visual analogue scale (VAS)) and overall health status (Euro Quality of Life-VAS (EQ-VAS)) were measured before and after 12 weeks.

DETAILED DESCRIPTION:
Main outcome:

The Perceived Stress Scale is a 10-item self report questionnaire that measures persons' evaluation of the stressfulness of the situations in the past month of their lives. The citation for the 10-item scale is Cohen, S., & Williamson, G. (1988). Perceived stress in a probability sample of the United States. In S. Spacapan & S. Oskamp (Eds.). The Perceived Stress Scale is the only empirically established index of general stress appraisal. "The PSS measures the degree to which situations in one's life are appraised as stressful" (Cohen, et al., 1983; p. 385).

PSS-10 scores are obtained by reversing the scores on the four positive items, e.g., 0=4, 1=3, 2=2, etc. and then summing across all 10 items. Items 4,5, 7, and 8 are the positively stated items. Scores can range from 0 to 40, with higher scores indicating greater stress.

The PSS is not a diagnostic instrument, so there are no cut-offs. There are only comparisons between people in a given sample. There are some normative data on the PSS based on a 1983 Harris Poll of a representative U.S. sample. These data may be helpful in providing comparisons, but they are over 20 years old. See: Cohen, S., & Williamson, G. (1988).

ELIGIBILITY:
Inclusion Criteria:

* The patients had sought treatment at the primary health centre during the previous 6 months.
* The stress-related symptoms included fatigue, insomnia, anxiety, depression, hypertension, and musculoskeletal discomfort in the neck and shoulders.

Exclusion Criteria:

* Inability to understand instructions, interpretation needs or physical or mental inability to carry out the Medical yoga exercises, such as mental retardation or dementia, and severe physical or mental illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2011-03; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Perceived stress scale | 12 week
  The Perceived Stress Scale is a 10-item self report questionnaire that measures persons' evaluation of the stressfulness of the situations in the past month of their lives. Cohen, S., & Williamson, G. (1988). PSS-10 scores are obtained by reversing the scores on the four positive items, e.g., 0=4, 1=3, 2=2, etc. and then summing across all 10 items. Items 4,5, 7, and 8 are the positively stated items. Scores can range from 0 to 40, with higher scores indicating greater stress.

SECONDARY OUTCOMES:
Shirom-Melamed Burnout Questionnaire | 12 week

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Westerdahl, PhD, Principal Investigator — Region Örebro County

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kohn M, Persson Lundholm U, Bryngelsson IL, Anderzen-Carlsson A, Westerdahl E. Medical yoga for patients with stress-related symptoms and diagnoses in primary health care: a randomized controlled trial. Evid Based Complement Alternat Med. 2013;2013:215348. doi: 10.1155/2013/215348. Epub 2013 Feb 26. PMID 23533465
- [Result] Anderzen-Carlsson A, Persson Lundholm U, Kohn M, Westerdahl E. Medical yoga: another way of being in the world-a phenomenological study from the perspective of persons suffering from stress-related symptoms. Int J Qual Stud Health Well-being. 2014 Jan 9;9:23033. doi: 10.3402/qhw.v9.23033. eCollection 2014. PMID 24434055